CLINICAL TRIAL: NCT01044641
Title: Measurement of Colloid Osmotic Pressure in Plasma and Interstitial Fluid in Children
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 065816
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Colloid Osmotic Pressure
Keywords: Colloid Osmotic pressure in interstitial fluid; Colloid Osmotic pressure in plasma; Protein fractions in interstitial fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interstitial fluid and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify normal values of colloid osmotic pressure in interstitial fluid and plasma in healthy children between 2 and 10 years.

DETAILED DESCRIPTION:
Measurements of colloid osmotic pressure (COP) by sampling of interstitial fluid from subcutaneous tissue and plasma are well documented in animal models and human adult studies. COP plays a major role in transcapillary fluid balance and is valuable in fluid therapy planning in critically ill patients. There are no data regarding interstitial fluid COP values in neither sick nor healthy children. Sampling of interstitial fluid by the wick method in children who is under general anaesthesia (ear-nose-throat operations) gives the opportunity to identify normal COP values in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 to 10 years

Exclusion Criteria:

* Medication
* Ongoing illness
* Syndromes

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Secondary care clinic (ENT)
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Colloid osmotic pressure | 60 minuttes after wick insertion

CONTACTS AND LOCATIONS:
Overall Officials: Hans Joergen T Guthe, MD, Principal Investigator — Hanukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

REFERENCES:
- [Derived] Guthe HJ, Indrebo M, Nedrebo T, Norgard G, Wiig H, Berg A. Interstitial fluid colloid osmotic pressure in healthy children. PLoS One. 2015 Apr 8;10(4):e0122779. doi: 10.1371/journal.pone.0122779. eCollection 2015. PMID 25853713